CLINICAL TRIAL: NCT05054062
Title: Sentinel Lymph Node Mapping With Superparamagnetic Iron Oxide for Melanoma: a Pilot Study in Healthy Participants to Establish an Optimal MRI Workflow Protocol
Brief Title: Sentinel Lymph Node Mapping Using Magtrace and MRI in Healthy Subjects for Potential Use in Melanoma Patients
Acronym: TRACIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Principal Investigator, James van Bastelaar, Head of department of Surgery (Surgical Oncologist), Zuyderland Medisch Centrum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METCZ20210103
Record Dates: First submitted 2021-09-09; First posted 2021-09-23 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Melanoma
Keywords: Magnetic tracer; Sentinel lymph node; Melanoma; MRI
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Healthy participants (Experimental)
  Interventions: Diagnostic Test: Sentinel node mapping using MRI

INTERVENTIONS:
Diagnostic Test: Sentinel node mapping using MRI — Sentinel lymph node mapping in melanoma patients using a magnetic tracer and MRI

SUMMARY:
Sentinel lymph node biopsy (SLNB) is crucial in the management of malignant melanoma treatment and is currently performed by pre-operatively inject a colloid nanomaterial labeled with Technetium (99mTc) as radioactive tracer. Intra-operatively, Patent Blue (PB) will be injected to improve the visualization of the lymphatic tract. However, current pre-operative SLN mapping technique, is associated with disadvantages as radiation exposure for both patients and health care personnel and logistic challenges, because of time constraints due to short half-live time of 99mTc.

Superparamagnetic iron oxide (SPIO) is novel, non-radioactive technique using a magnetic tracer (Magtrace® (Endomagnetics Ltd.)) and several studies showed that SPIO is non-inferior to dual tracing with 99mTc and PB in breast cancer patients. SPIO is expected to be non-inferior to dual tracing with 99mTc and PB in melanoma patients. However, further research is needed to demonstrate the use of SPIO in pre-operative Magnetic Resonance Imaging (MRI) scanning. Guidance on pre-operative MRI use is rather limited, though fundamental in the intended research process.

Hence, the aim of this subprotocol study, which includes healthy subjects, is to develop a pre-operative MRI protocol for melanoma patients. The acquired knowledge will be used to design a feasibility study, including a larger group of melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants;
* Participants should be ≥18 years of age at the time of consent;
* Participants should be willing to provide informed consent.

Exclusion Criteria:

* Known intolerance/hypersensitivity to iron, dextran compounds or Magtrace® itself;
* Standard MRI exclusion criteria:
* Implantable (electrical) devices (e.g. pacemaker, cochlear implants, neurostimulator);
* Any other metal implants;
* Claustrophobia;
* MR-incompatible prosthetic heart valves;
* Tattoos inked with metallic dye.
* Participants who refuse to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-08-20 (Actual)

PRIMARY OUTCOMES:
SPIO dosage in milliliters | Three weeks
  SPIO dosage in milliliters will be assessed to develop a pre-operative MRI protocol. Testing will be perform in healthy subjects.
Massage duration in seconds | Three weeks
  Massage duration in seconds will be assessed to develop a pre-operative MRI protocol. Testing will be perform in healthy subjects.
Time to artefact appearance in minutes | Three weeks
  Time to artefact appearance in minutes will be assessed to develop a pre-operative MRI protocol. Testing will be perform in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aldenhoven L, Frotscher C, Korver-Steeman R, Martens MH, Kuburic D, Janssen A, Beets GL, van Bastelaar J. Sentinel lymph node mapping with superparamagnetic iron oxide for melanoma: a pilot study in healthy participants to establish an optimal MRI workflow protocol. BMC Cancer. 2022 Oct 14;22(1):1062. doi: 10.1186/s12885-022-10146-w. PMID 36241982